CLINICAL TRIAL: NCT03998449
Title: Evaluation of Immunogenicity of Cholera Vaccine in Children With Inflammatory Bowel Disease
Brief Title: Immunogenicity of Cholera Vaccine in Children With IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Lukasz Dembinski, Principal Investigator, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Dembinski2019
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Cholera; Inflammatory Bowel Diseases
MeSH Terms: conditions — Cholera; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cholera vaccination (Experimental): Two doses of the vaccine against cholera
  Interventions: Biological: Vaccination against cholera

INTERVENTIONS:
Biological: Vaccination against cholera — Participants will receive two doses of an oral cholera vaccine with an interval of 2-4 weeks.

SUMMARY:
Assessment of the immunogenicity and safety of immunization against cholera in children with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Crohn's disease or ulcerative colitis based on standard clinical, endoscopic, histologic and radiographic criteria (Porto criteria),
* no vaccination against cholera in the past,
* written consent of the patient's legal guardians and the patient himself if he/she turns 16 years of age.

Exclusion Criteria:

* serious exacerbation of inflammatory bowel disease defined as Paediatric Ulcerative Colitis Activity Index (PUCAI) > 65 points for patients with ulcerative colitis or Pediatric Crohn's Disease Activity Index (PCDAI) > 40 points for patients with Crohn's disease.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Achieving seroprotective antibody concentration | 4-6 weeks after the second dose
  Serum antibody concentration indicating protection against cholera.

SECONDARY OUTCOMES:
Adverse effects | 3 days after each dose
  Evaluation of adverse effects after vaccination.
Inflammatory bowel disease exacerbation occurrence. | 4-6 weeks after the second dose
  Disease exacerbation assessed according to the Paediatric Ulcerative Colitis Activity Index (PUCAI) for patients with ulcerative colitis or Pediatric Crohn's Disease Activity Index (PCDAI) for patients with Crohn's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Banaszkiewicz, MD, PhD, Study Director — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No